CLINICAL TRIAL: NCT01852214
Title: A Pharmacodynamic Comparison of Prasugrel vs. Ticagrelor in Patients With Type 2 Diabetes Mellitus and Coronary Artery Disease
Brief Title: Pharmacodynamic Effect of Prasugrel vs. Ticagrelor in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UFJ 2011-184
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease
Keywords: Diabetes mellitus; Coronary artery disease; prasugrel; ticagrelor
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel first, then ticagrelor (Active Comparator): Patients randomized to prasugrel will receive prasugrel loading dose followed by maintenance dose. Randomized treatment will be maintained for 1-week (7±2 days). After completion of the 1-week treatment period, patients will discontinued the study medications for 2-4 weeks (wash-out period) and then will cross over to the alternate treatment (ticagrelor), which will be administered for 1-week.
  Interventions: Drug: Prasugrel; Drug: Ticagrelor
- Ticagrelor first, then prasugrel (Active Comparator): Patients randomized to ticagrelor will receive prasugrel loading dose followed by maintenance dose. Randomized treatment will be maintained for 1-week (7±2 days). After completion of the 1-week treatment period, patients will discontinued the study medications for 2-4 weeks (wash-out period) and then will cross over to the alternate treatment (prasugrel), which will be administered for 1-week.
  Interventions: Drug: Prasugrel; Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Patients receiving prasugrel will be treated with 60mg loading dose and 10mg maintenance dose
  Other Names: Effient
Drug: Ticagrelor — Patients receiving ticagrelor will be treated with a 180mg loading dose and 90mg bid maintenance dose
  Other Names: Brillinta

SUMMARY:
Patients with diabetes mellitus (DM) have an increased risk of adverse atherothrombotic events. This may be in part attributed to the fact that these patients have reduced response to oral antiplatelet medications, in particular the P2Y12 receptor inhibitor clopidogrel, used for secondary prevention of ischemic events. Prasugrel and ticagrelor are recently approved P2Y12 receptor inhibitors which, compared with clopidogrel, have more potent antiplatelet effects. Head-to-head comparisons between the two drugs are lacking.

DETAILED DESCRIPTION:
Patients with diabetes mellitus (DM) have an increased risk of adverse atherothrombotic events. This may be in part attributed to the fact that these patients have reduced response to oral antiplatelet medications, in particular the P2Y12 receptor inhibitor clopidogrel, used for secondary prevention of ischemic events. Upregulation of platelet P2Y12 receptor mediated signaling has been shown in DM patients and may contribute to these pharmacodynamic observations, suggesting the need for more potent P2Y12 inhibiting strategies in these patients. Prasugrel and ticagrelor are recently approved P2Y12 receptor inhibitors which, compared with clopidogrel, have more potent antiplatelet effects. Therefore, prasugrel and ticagrelor represent attractive treatment options for patients with DM. This is also supported by the DM sub-group analysis of the pivotal TRITON-TIMI 38 (Trial to Assess Improvement in Therapeutic Outcomes by Optimizing Platelet Inhibition with Prasugrel-Thrombolysis in Myocardial Infarction) and PLATO (Platelet Inhibition and Patient Outcomes) trials, which have led to approval of prasugrel and ticagrelor, respectively. Although results of these sub-group analysis suggest that prasugrel is associated with an enhanced benefit in DM patients, while ticagrelor effects in DM patients are consistent with the overall study population, only head-to-head comparisons between the two drugs can elucidate if these exert differential effects on platelets from DM patients. However, the pharmacodynamic studies comparing prasugrel with ticagrelor in DM patients are lacking. The ever growing DM population at high risk of recurrent atherothrombotic events underscores the need to define antiplatelet treatment strategies leading to more optimal platelet inhibition in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known (angiographically documented) CAD.
* On maintenance treatment with aspirin (81 mg per day) for at least 1-month as per standard of care.
* Type 2 DM on treatment with oral hypoglycemic agents and/or insulin.
* Age between 18 and 74 years old.

Exclusion Criteria:

* History of stroke, transient ischemic attack or intracranial bleeding.
* On treatment with a P2Y12 receptor antagonist (ticlopidine, clopidogrel, prasugrel, ticagrelor).
* Known allergies to aspirin, ticlopidine, clopidogrel, prasugrel, ticagrelor.
* Weight <60kg.
* On treatment with oral anticoagulant (Vitamin K antagonists, dabigatran).
* Blood dyscrasia or bleeding diathesis.
* Platelet count <80x106/mL.
* Hemoglobin <10 g/dL.
* Active bleeding or hemodynamic instability.
* Creatinine Clearance <30 mL/minute.
* Baseline ALT >2.5 times the upper limit of normal.
* Hb A1c ≥ 10 mg/dL within 3 months.
* Patients with sick sinus syndrome (SSS) or high degree AV block without pacemaker protection.
* Drugs interfering CYP3A4 metabolism (to avoid interaction with Ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromizycin.
* Pregnant females*.

  * Women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franchi F, Rollini F, Aggarwal N, Hu J, Kureti M, Durairaj A, Duarte VE, Cho JR, Been L, Zenni MM, Bass TA, Angiolillo DJ. Pharmacodynamic Comparison of Prasugrel Versus Ticagrelor in Patients With Type 2 Diabetes Mellitus and Coronary Artery Disease: The OPTIMUS (Optimizing Antiplatelet Therapy in Diabetes Mellitus)-4 Study. Circulation. 2016 Sep 13;134(11):780-92. doi: 10.1161/CIRCULATIONAHA.116.023402. Epub 2016 Aug 24. PMID 27559041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2013 and July 2015, a total of 61 subjects agreed to participate in the study; 11 subjects were excluded and thus a total of 50 subjects were randomized (prasugrel first n=26; ticagrelor first n=24).
Pre-assignment Details: 11 subjects were excluded before randomization: withdrawn of consent (n=4), screen failure (n=4), unable to draw blood (n=3).
Groups:
- Prasugrel First, Then Ticagrelor: Prasugrel: Patients randomized to prasugrel will be treated with 60mg loading dose and 10mg maintenance dose
  Ticagrelor: Patients randomized to ticagrelor will be treated with a 180mg loading dose and 90mg bid maintenance dose
- Ticagrelor First, Then Prasugrel: Ticagrelor: Patients randomized to ticagrelor will be treated with a 180mg loading dose and 90mg bid maintenance dose
  Prasugrel: Patients randomized to prasugrel will be treated with 60mg loading dose and 10mg maintenance dose
Period: Period 1
Arm/Group | Prasugrel First, Then Ticagrelor | Ticagrelor First, Then Prasugrel
Started | 26 | 24
Completed | 25 | 21
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout Period
Arm/Group | Prasugrel First, Then Ticagrelor | Ticagrelor First, Then Prasugrel
Started | 25 | 21
Completed | 25 | 20
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Prasugrel First, Then Ticagrelor | Ticagrelor First, Then Prasugrel
Started | 25 | 20
Completed | 25 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All analyses of platelet function were conducted on the pharmacodynamic population, which was defined as all randomized subjects who received study drug, successfully completed at least one treatment period of the study and had valid data for the primary end point (n=46)
Groups:
- Overall Population: Subjects with type 2 diabetes mellitus and coronary artery disease
Arm/Group | Overall Population
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Type of diabetes [Number; unit: participants]
  Insulin-dependent | 26
  Non-insulin-dependent | 20

OUTCOME MEASURES:

1. Primary Outcome: P2Y12 Reaction Units
Description: The primary endpoint is the comparison of the P2Y12 reaction units (PRU) values determined by VerifyNow between both treatments (ticagrelor or prasugrel). Treatment effects were evaluated comparing PRU observed in the overall patient population after prasugrel treatment with those achieved after ticagrelor regardless of the sequence.
Time Frame: 1 week
Population: All analyses of platelet function conducted on all randomized subjects who received study drug, successfully completed at least one treatment period of the study and had valid data for the primary end point.
Measure: Least Squares Mean (95% Confidence Interval); unit: PRU
Groups:
- Prasugrel: Patients received 60mg loading dose and 10mg maintenance dose
- Ticagrelor: Patients received a 180mg loading dose and 90mg bid maintenance dose
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 45 | 46
PRU | 83 [63 to 103] | 52 [32 to 72]
Statistical Analysis 1: Comparison: Prasugrel vs Ticagrelor; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis

2. Secondary Outcome: P2Y12 Reaction Units
Description: Comparison of the P2Y12 reaction units (PRU) values determined by VerifyNow between both treatments (ticagrelor or prasugrel)
Time Frame: 2 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: PRU
Groups:
- Ticagrelor: Patients received 180mg loading dose and 90mg bid maintenance dose
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 45 | 46
PRU | 97 [78 to 117] | 75 [56 to 95]
Statistical Analysis 1: Comparison: Prasugrel vs Ticagrelor; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis

3. Secondary Outcome: Platelet Reactivity Index
Description: The comparison of the platelet reactivity index (PRI) values determined by vasodilator-stimulated phosphoprotein (VASP) between both treatments (ticagrelor or prasugrel). VASP was measured by quantitative flow cytometry using commercially available labelled monoclonal antibodies. A low PRI is indicative of high platelet inhibition.
Time Frame: 1 week
Measure: Least Squares Mean (95% Confidence Interval); unit: PRI
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 45 | 46
PRI | 36 [30 to 41] | 36 [30 to 42]

4. Secondary Outcome: Platelet Reactivity Index
Description: as for outcome 3
Time Frame: 2 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: PRI
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 45 | 46
PRI | 35 [25 to 45] | 37 [29 to 46]

ADVERSE EVENTS:
Time Frame: Through study completion, up to 46 days.
Groups:
- Safety Population: Patients Receiving Prasugrel; Safety Population: Patients Receiving Ticagrelor: Safety analyses were conducted on the safety population, which included all patients exposed to at least one dose of the study drug, and are reported according to the intervention received at the time the adverse event occurred.
Arm/Group | Safety Population: Patients Receiving Prasugrel | Safety Population: Patients Receiving Ticagrelor
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/49
Other Adverse Events (participants affected / at risk) | 4/46 | 10/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population: Patients Receiving Prasugrel (N=46) | Safety Population: Patients Receiving Ticagrelor (N=49)
BARC type 1 bleeding (Blood and lymphatic system disorders) | 1 | 1 — Bleeding events were classified according to the BARC (Bleeding Academic Research Consortium) definition
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No